CLINICAL TRIAL: NCT02918630
Title: E-cigarettes to Promote Smoking Reduction Among Individuals With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jin Ho Yoon, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-16-0667
Record Dates: First submitted 2016-09-20; First posted 2016-09-29 (Estimated); Results first posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-06

CONDITIONS: Tobacco Smoking
Keywords: E-cigarettes; Schizophrenia
MeSH Terms: conditions — Tobacco Smoking; Vaping; Schizophrenia | interventions — Tobacco Use Cessation Devices; Electronic Nicotine Delivery Systems

ARMS (2):
- Nicotine Replacement Therapy - Nicotine Patch (Active Comparator): Participants will receive nicotine patch (21 mg) starting study Week 1. Participants will be instructed to apply a new patch each morning.
  Interventions: Drug: Nicotine Patch
- Nicotine Replacement Therapy + E-cigarette (Experimental): The e-cigarette will consist of 1) a 3.3 V, 1000 mAh battery; and 2) a 1.5 Ohm, dual-coil cartomizer (SmokTech; Shenzhen, China). Study staff will load the cartomizer with 1 ml tobacco flavored 70% propylene glycol/30% vegetable glycerin liquid containing nicotine concentrations 36 mg/ml (AVAIL; Richmond, Virginia, USA).
  Interventions: Drug: Nicotine Patch; Drug: E-cigarette

INTERVENTIONS:
Drug: Nicotine Patch — Participants will receive nicotine patch (21 mg) starting study Week 1. Participants will be instructed to apply a new patch each morning.
Drug: E-cigarette — The e-cigarette will consist of 1) a 3.3 V, 1000 mAh battery; and 2) a 1.5 Ohm, dual-coil cartomizer (SmokTech; Shenzhen, China). Study staff will load the cartomizer with 1 ml tobacco flavored 70% propylene glycol/30% vegetable glycerin liquid containing nicotine concentrations 36 mg/ml (AVAIL; Richmond, Virginia, USA).
  Arms: Nicotine Replacement Therapy + E-cigarette

SUMMARY:
The purpose of this study is to assess if access to an electronic nicotine delivery device, or e-cigarette, in addition to nicotine patch (21 mg) can help reduce cigarette smoking among individuals diagnosed with schizophrenia compared to nicotine patch alone.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with schizophrenia
* Be in stable medical condition (DSM-V)
* report smoking ≥10 tobacco cigarettes/day
* present a breath CO ≥10 ppm
* report wanting to reduce their cigarette smoking
* be fluent in English
* have a stable living situation

Exclusion Criteria:

* be currently pregnant or breastfeeding
* report wanting to quit smoking in the immediate future
* test positive for illicit drugs except THC
* have any illness, medical condition, or use of medications, which in the opinion of the study physicians would preclude safe and/or successful completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-10; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Ho Yoon, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nicotine Replacement Therapy - Nicotine Patch | Nicotine Replacement Therapy + E-cigarette
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine Replacement Therapy - Nicotine Patch | Nicotine Replacement Therapy + E-cigarette | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (4.377) | 44.6 (1.2) | 48.3 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Smoking as Assessed by Breath Carbon Monoxide Levels
Time Frame: Baseline, Week 5
Measure: Mean (Standard Deviation); unit: parts per million (ppm)
Arm/Group | Nicotine Replacement Therapy - Nicotine Patch | Nicotine Replacement Therapy + E-cigarette
Number analyzed (Participants) | 4 | 3
parts per million (ppm) | -18 (24) | -4.3 (3.1)

2. Primary Outcome: Change in Smoking as Assessed by Urinary Cotinine Levels
Time Frame: Baseline, Week 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nicotine Replacement Therapy - Nicotine Patch | Nicotine Replacement Therapy + E-cigarette
Number analyzed (Participants) | 4 | 3
ng/mL | 0 (0) | 0 (0)

3. Primary Outcome: Number of Cigarettes Smoked Per Day as Assessed by Self-report Via Timeline Follow-back
Description: Timeline follow-back involves asking participants to retrospectively estimate their cigarette use in the week prior to the interview date. An average number of cigarettes per day was calculated for each participant, and the average of the average number of cigarettes per day for all participants is reported below.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: number of cigarettes per day
Arm/Group | Nicotine Replacement Therapy - Nicotine Patch | Nicotine Replacement Therapy + E-cigarette
Number analyzed (Participants) | 4 | 3
number of cigarettes per day | 13 (6) | 23 (16)

4. Secondary Outcome: Feasibility as Assessed by Percent of Participants Who Completed the Study
Time Frame: week 5
Measure: Number; unit: percent of participants
Arm/Group | Nicotine Replacement Therapy - Nicotine Patch | Nicotine Replacement Therapy + E-cigarette
Number analyzed (Participants) | 4 | 3
percent of participants | 100 | 100

5. Primary Outcome: Number of Cigarettes Smoked Per Day as Assessed by Self-report Via Timeline Follow-back
Description: as for outcome 3
Time Frame: week 5
Measure: Mean (Standard Deviation); unit: number of cigarettes per day
Arm/Group | Nicotine Replacement Therapy - Nicotine Patch | Nicotine Replacement Therapy + E-cigarette
Number analyzed (Participants) | 4 | 3
number of cigarettes per day | 9 (7) | 12 (7)

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Nicotine Replacement Therapy - Nicotine Patch | Nicotine Replacement Therapy + E-cigarette
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Replacement Therapy - Nicotine Patch (N=4) | Nicotine Replacement Therapy + E-cigarette (N=3)
Drowsiness (General disorders) | 4 (4) | 3 (3)
Not sleeping well (General disorders) | 2 (2) | 3 (3)
Headache (General disorders) | 3 (3) | 3 (3)
Nervousness (Psychiatric disorders) | 3 (3) | 3 (3)
Blurry vision (Eye disorders) | 3 (3) | 3 (3)
Dizziness (General disorders) | 3 (3) | 3 (3)
Tremor (shaky hands) (General disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Stomach pain (cramps) (General disorders) | 4 (4) | 3 (3)
Muscle aches (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Heart racing (Cardiac disorders) | 3 (3) | 3 (3)
Chest pain (General disorders) | 3 (3) | 3 (3)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Increased urination (Renal and urinary disorders) | 3 (3) | 3 (3)
Change in sexual function (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Weakness (General disorders) | 4 (4) | 3 (3)
Sweating (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Dry mouth (General disorders) | 4 (4) | 3 (3)
Fatigue (General disorders) | 3 (3) | 3 (3)
Difficulty walking (General disorders) | 3 (3) | 2 (2)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Swelling (General disorders) | 2 (2) | 2 (2)
Fever/chills (General disorders) | 0 (0) | 1 (1)
Loss of appetite (General disorders) | 3 (3) | 2 (2)
Confusion (General disorders) | 3 (3) | 1 (1)
Cloudiness (General disorders) | 3 (3) | 2 (2)
Memory loss (General disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT02918630/Prot_SAP_000.pdf